CLINICAL TRIAL: NCT06511869
Title: A Phase II, Open-Label, Multicenter Study to Assess the Safety and Anti-Tumor Efficacy of AZD4205 in Participants With Peripheral T Cell Lymphoma Who Have Responded After First-Line Standard Therapy
Brief Title: AZD4205 in Peripheral T Cell Lymphoma Following First-Line Therapy (JACKPOT26)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2021J0005
Record Dates: First submitted 2024-07-15; First posted 2024-07-22 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD4205 treatment (Experimental): Cohort 1: Participants achieving a CR as assessed by the investigator according to Lugano criteria following the first-line systemic therapy.
  Cohort 2: Participants achieving a PR as assessed by the investigator according to Lugano criteria following the first-line systemic therapy.
  Interventions: Drug: AZD4205

INTERVENTIONS:
Drug: AZD4205 — AZD4205 capsules administered at 150 mg orally, once daily, in 28-day cycle.

SUMMARY:
This study is intended to assess the safety and anti-tumor activity of AZD4205 at 150 mg once daily in participants with PTCL who have achieved tumor response after first-line systemic therapy (with or without combination radiotherapy) and are ineligible for HSCT assessed by the investigator as ineligible for HSCT or have no plan for HSCT.

ELIGIBILITY:
Inclusion criteria

1. ≥ 18 years old.
2. ECOG status score ranging from 0 to 1, without any deterioration in the past two weeks.
3. Life expectancy ≥ 3 months.
4. Have histopathologically confirmed PTCL that meets the pathological subtypes (except for ALCL-ALK+) as specified in the latest WHO classification of lymphoid neoplasms in 2016.
5. Must be assessed to achieve complete or partial response according to Lugano's criteria after first-line systemic standard of therapy:

   * The participants should be assessed as ineligible for HSCT
   * For participants with CR, the end of initial treatment should be ≤ 3 months from the planned first dose in this study.
6. Adequate bone marrow hematopoietic function and organ function reserve.
7. LVEF ≥ 50% by ECHO.
8. Should be able to follow the relevant requirements of this study for medication and follow-up.
9. If there is a potential for conception for the female spouses (partners) of male participants, the spouses (partners) should take physical contraceptive measures (such as condoms) during the participant participating in the trial and within 6 months after the end of treatment.
10. Male participants should also avoid sperm donation during the trial and within 6 months after the end of treatment.
11. Female participants should take adequate contraceptive measures and vasoligation of the partner during the trial and within 3 months after the end of the trial. All hormonal contraceptive methods (except abstinence) should be used in conjunction with the use of a condom by the male partner. Breastfeeding is prohibited for female participants. Female participants of conception potential should have a negative pregnancy test prior to initiation of treatment.

Exclusion criteria

1. With any of the following treatment history:

   * The use of the investigational product or investigational product in another project within 30 days prior to the start of dosing in this study.
   * The cytotoxic chemotherapeutic agents are not discontinued within 21 days prior to the start of dosing in this study.
   * Prior use of histone deacetylase (HDAC) inhibitors (e.g., romidepsin, chidamide, belinostat) or pralatrexate within 1 week prior to the start of dosing in this study.
   * Prior use of corticosteroid therapy at equivalent prednisone dose > 15 mg/day within 1 week prior to the start of dosing in this study.
   * Undergoing major surgery (excluding vascular access surgery) or serious trauma within 4 weeks prior to the start of dosing in this study; or anticipated to undergo potential surgery after the start of dosing in this study.
   * Prior use of anti-tumor macromolecular antibody agents (including brentuximab vedotin) within 4 weeks; radiation therapy within 3 weeks; and other toxin/isotope-immune antibody couplers within 10 weeks prior to the start of dosing in this study.
   * With prior use of JAK or STAT3 inhibitors.
   * Prior use of anti-tumor immunotherapy (e.g., immune checkpoint inhibitors, including PD-1, PD-L1, and CTLA-4) within 28 days prior to the start of dosing in this study. For participants treated with other types of novel therapy, whether they can be included may be jointly decided by the investigator and the sponsor's study physician.
   * Vaccination with attenuated vaccines or viral vector vaccines within 28 days prior to the start of dosing in this study.
   * Currently on treatment with vitamin K antagonists, antiplatelets, and anticoagulants (or these drugs cannot be discontinued within 1 week prior to the start of dosing in this study).
   * Currently on treatment with (or unable to discontinue the use within 1 week prior to the start of dosing in this study) certain known drugs, herbs, or supplements that may significantly induce or inhibit CYP3A or can serve as sensitive substrates of BCRP/P-gp, with low therapeutic indexes.
2. With unresolved > CTCAE Grade 1 adverse drug reactions (except alopecia) prior to the start of dosing in this study.
3. Central nervous system or meninges involvement by the lymphoma.
4. With significant lung function impairment (i.e., pulmonary function tests show FEV1 and DLCO < 60% of predicted values). Participants with prior history of non-infectious pneumonitis, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy, or evidence showing clinically active interstitial lung disease.
5. With diseases or conditions requiring treatment with immunosuppressive agents, similar biological agents, or non-steroidal analgesic-antipyretic drugs.
6. Active infection, including:

   * Known active/latent tuberculosis (screening should be performed according to the routine procedures of local clinical sites, such as PPD test, T-SPOT, and X-ray/CT).
   * With positive HIV test or serological hepatitis markers.
   * Active viral infections (e.g., herpes zoster) other than hepatitis B or hepatitis C.
   * Infections requiring oral or intravenous antimicrobial therapy.
   * Bacterial infection within 30 days, including pneumonia.
7. Any of the following cardiac abnormalities:

   * With congestive heart failure (CHF) > NYHA Class II.
   * With significant clinical manifestations of valvular disease and hypertrophic/constrictive cardiomyopathy.
   * With serious cardiac rhythm, conduction, morphological abnormalities on any resting ECG, such as complete left bundle branch block, 2/3-degree atrioventricular block, and PR interval > 250 ms.
   * Ventricular arrhythmia requiring treatment.
   * Acute myocardial infarction (AMI) within 6 months prior to the start of treatment in the trial; unstable angina pectoris or new angina pectoris.
   * Who have undergone heart transplantation.
   * Corrected QTcF interval (QTc) > 450 ms on resting ECG at screening.
   * With increased risks of QT prolongation or arrhythmia (e.g., heart failure, hypokalemia, congenital long QT syndrome, or taking other drugs causing QT prolongation; or with a family history of long QT syndrome; or those with first-degree relatives showing unexpected sudden death under 40 years of age.
   * Prior or current history of thrombotic diseases such as pulmonary embolism and deep vein thrombosis.
8. Prior history of malignancies (except completely eradicated cervical, uterine, basal cell, or squamous cell carcinoma in situ, or non-melanoma skin carcinoma in situ) within 5 years prior to enrollment.
9. With symptoms of intractable nausea or vomiting that cannot be well controlled with supportive treatment, chronic gastrointestinal disease, capsule dysphagia, or prior surgical removal of bowel segments that may compromise adequate absorption of the drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events (graded by CTCAE version 5.0) | up to 2 years
  To assess the safety and tolerability of AZD4205 as maintenance/consolidation therapy in PTCL participants achieving tumor response after first-line systemic therapy

SECONDARY OUTCOMES:
Cohort 1: Disease Free Survival (DFS) | up to 2 years
  To assess the anti-tumor activity of AZD4205 as maintenance/consolidation therapy in PTCL participants achieving tumor response after first-line systemic therapy
Cohort 1: Disease Free Survival (DFS) rate at 1 year from the first dose of investigational product | 1 year
  To assess the anti-tumor activity of AZD4205 as maintenance/consolidation therapy in PTCL participants achieving tumor response after first-line systemic therapy
Cohort 2: Objective Response Rate (ORR) | up to 2 years
  To assess the anti-tumor activity of AZD4205 as maintenance/consolidation therapy in PTCL participants achieving tumor response after first-line systemic therapy
Cohort 2: Duration of Response (DoR) | up to 2 years
  To assess the anti-tumor activity of AZD4205 as maintenance/consolidation therapy in PTCL participants achieving tumor response after first-line systemic therapy
Cohort 2: Progression-free Survival (PFS) | up to 2 years
  To assess the anti-tumor activity of AZD4205 as maintenance/consolidation therapy in PTCL participants achieving tumor response after first-line systemic therapy
Cohort 2: Progression-free Survival (PFS) rate at 1 year from the first dose of investigational product | 1 year
  To assess the anti-tumor activity of AZD4205 as maintenance/consolidation therapy in PTCL participants achieving tumor response after first-line systemic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (23):
- China (23):
  - Anhui Provincial Hospital (The First Affiliated Hospital of USTC), Hefei, Anhui
  - Peking university Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Research Center of Clinical Trials, The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shandong Cancer Hospital & Institution, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No